CLINICAL TRIAL: NCT06882486
Title: Post-immunotherapy Nephrectomy for Metastatic Kidney Cancer After Complete or Major Response to Systemic Therapy
Acronym: NAMECAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAMECAR-IPC 2024-054
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Nephrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nephrectomy (Experimental): delayed nephrectomy and discontinuation of systemic treatment
  Interventions: Procedure: nephrectomy
- no nephrectomy (No Intervention): no nephrectomy and continuation of systemic treatment

INTERVENTIONS:
Procedure: nephrectomy — Nephrectomy scheduled within 3 months of inclusion. Patients may continue their systemic treatment at the usual rate until D-5 prior to surgery. Treatment will not be resumed after surgery. Surgery may consist of partial or enlarged nephrectomy, with or without associated lymph node dissection, depending on technical possibilities and at the surgeon's discretion.
  Arms: nephrectomy

SUMMARY:
In the current era of immune checkpoint inhibitors (ICI), the role and timing of nephrectomy remains unknown, particularly in cases of residual kidney disease after a major response at metastatic sites. In these cases, the rationale for a delayed nephrectomy is that it might achieve a long-term response. This strategy could allow some patients to discontinue treatment and maintain tumor response. Furthermore, this approach might provide a potentially curative option for patients with metastases that are managed with and responding to ICI.

Regarding the results of our first retrospective cohort data (showing that two thirds of patients are free from recurrence without systemic treatment after nephrectomy), we designed a non-comparative randomized phase II trial assessing progression-free survival of patients with complete response or major partial response after ICI-based treatment, operated on delayed nephrectomy with discontinuation of systemic therapy (experimental arm) and in patients managed with continuation of systemic therapy without nephrectomy (control arm).

In a de-escalation approach, this strategy may have sense to allow patients with an excellent response to immunotherapy to stop systemic treatment with a curative objective and a substantial impact from a medico-economic point of view.

DETAILED DESCRIPTION:
Patients with metastatic kidney cancer will be treated according to current first-line treatment guidelines.

Patients may be included in the study (by signing a consent form) and randomized if a complete response (CR) or metastatic partial response (mPR) (>75%) is achieved with immunotherapy-based systemic therapy.

In the centers participating in the ancillary study, patients in the experimental arm (arm A) will undergo renal MRI and PSMA PET (positron emission tomography) scan prior to nephrectomy.

Arm A patients will undergo nephrectomy (partial or enlarged, depending on technical possibilities and surgeon's discretion), after which systemic treatment will be discontinued.

Patients in arm B will not undergo surgery, and will continue their systemic treatment unchanged (interrupted in the event of toxicity, in accordance with current recommendations).

In both arms, follow-up will consist of a biological and CT scan evaluation every 3 months for 2 years.

The primary objective is to evaluate the efficacy of the experimental strategy in terms of progression-free survival, progression being defined according to the usual RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged ≥ 18 years
2. Diagnosed with synchronous metastatic kidney cancer
3. With primary tumor still in place (no primary cytoreductive nephrectomy)
4. Having received systemic ICI immunotherapy-based combination therapy
5. In CR or mPR (defined as >75% response in metastatic lesions from baseline) according to the Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1), excluding the primary renal lesion.
6. Signed consent to participate
7. Affiliated to the national social security scheme or beneficiaries of such a scheme

Exclusion Criteria:

1. Women who are or may become pregnant (without effective contraception) or who are breast-feeding.
2. Person in an emergency situation or unable to give consent.
3. An adult under legal protection (guardianship, curators or safeguard of justice),
4. Inability to undergo medical follow-up for geographical, social or psychological reasons.
5. Patients who have undergone prior cytoreductive nephrectomy
6. Patients considering nephrectomy for symptomatic disease, but without major response (CR or mPR) in metastatic disease
7. Patients with non-metastatic disease at diagnosis who have received ICI in a neo-adjuvant setting
8. Patients with contraindications to surgery or ineligible for nephrectomy
9. Patients not wishing to undergo nephrectomy
10. Patients with end-stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 24 month
  post-randomization progression-free survival

SECONDARY OUTCOMES:
Overall survival | 24 month
  Overall post-randomization survival
Intraoperative and postoperative complications | 30 days
  Rate of intraoperative and postoperative complications
Immunotherapy-related adverse events | 24 months
  Rate of immunotherapy-related adverse events (including CTCAE grade ≥ 3)